CLINICAL TRIAL: NCT03649854
Title: Measurement of Tricuspid Annular Plane Systolic Excursion in Transesophageal Echocardiography Using Two Deep Transgastric Views
Brief Title: Measurement of Tricuspid AnnularPlane Systolic Excursion in Transesophageal Echocardiography
Acronym: TAPSE
Status: Completed | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Anaesthesia, Principal Investigator, National University Hospital, Singapore
Other Study IDs: 2014/00576
Record Dates: First submitted 2018-08-23; First posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Right Heart Dysfunction
Keywords: TAPSE; Right heart function

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to measure TAPSE in TEE using two deep transgastric views. This is a prospective comparative diagnostic study where 21 CABG patients who are enrolled for the study will be studied during the intraoperative period. The choice of general anaesthesia, hemodynamic management will be at the discretion of the anaesthesiologist in charge of the patient. The monitoring technique is standard as per any cardiac surgery with cardiopulmonary bypass. After induction of anaesthesia, TEE probe will be inserted by the PI or the Co-Investigator and the required TEE standard views and deep TG view of the right heart at zero degree and Deep TG view at 100-150 degrees will be acquired TAPSE will be measured in both the views using Mmode.

The measurement will be done as follows: After acquiring the deep TG views the M mode cursor is aligned with the longitudinal motion the lateral tricuspid annulus. Once the Mmode picks up a good signal, 3 cycles are chosen and measured using calipers, and an average reading is taken. TAPSE will be used to evaluate the right heart function during the intraoperative period so that the patients with deteriorating right heart function can be identified and treatment started early. The potential benefits include the simplicity and reproducibility of the technique.

DETAILED DESCRIPTION:
Right ventricular failure(RVF) is an important cause of postoperative morbidity and mortality after cardiac surgery. Severe refractory RVF requiring prolonged inotropic support or RV assist device occurs in approximately 0.1% of patients after cardiotomy and in 20-30% of patients after left ventricular failure. The survival rate in these patients may be as low as 25 to 30%. Early diagnosis and prompt instituition of therapy may improve survival. In the intraoperative setting TEE is becoming the mainstay in the assessment of right ventricular function. However, presently it is not systematic and objective assessment of RV is not uniformly carried out. This is partly due to the enormous attention given to the evaluation of the left ventricle and the echo challenges of right heart imaging during intraoperative period.

In 2010 the ASE released the guidelines on Right heart. It recommends Fractional Area change, Tricuspid Annular Plane Systolic Excursion(TAPSE) and Peak Systolic tissue velocity of tricuspid annulus as simple reproducible measurements that can be done in all the patients. The guidelines are based on Transthoracic Echocardiography measurements. The Transesophageal echocardiography which is used during cardiac surgery poses unique challenges when assessing the right heart. The right ventricle lies in the far field where the resolution is not good, and is made worse by the extensive apical trabeculations ; these factors make endocardial border tracing difficult. In addition, the tissue Doppler and M mode alignment of the tricuspid annulus is not possible in the mid oesophageal views. Recently, a deep trans gastric view more than 120-150 degrees has been suggested by Denault et al which would give an alignment for tissue and pulse wave Doppler but TAPSE hasn't been studied using this view. The investigators have found a novel Deep trans gastric right heart view at zero degrees , which provides a good alignment for Doppler and M mode from which TAPSE, Peak systolic tissue velocity of the Tricuspid annulus, and Right ventricular performance index can be readily measured. We believe that this single view which can be easily acquired in most patients can comprehensively assess the systolic and diastolic function of the right heart during the intraoperative period.

The investigators propose that TAPSE can be accurately measured using M mode in the deep transgastric right heart view at zero degrees because it provides perfect alignment with longitudinal excursion of the lateral tricuspid annulus. Since the frame rate of M mode is very high, distance can be more accurately measured than any other technique.

The aim of this study is to compare TAPSE measurement using Mmode in the two Deep transgastric views: Deep TG view at 120- 150 degrees

ELIGIBILITY:
Inclusion Criteria:

* Ejection fraction greater than 40% No other valvular involvement other than mild mitral regurgitation

Exclusion Criteria:

* Hemodynamically unstable patients
* Intubated and sedated patients
* Emergency patients from cath lab

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for coronary artery bypass surgery at National university hospital are included in the study
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2014-08-15 (Actual); Primary Completion 2015-03-23 (Actual); Study Completion 2015-08-14 (Actual)

PRIMARY OUTCOMES:
New method for assessing right heart function | During systole intraoperatively
  TAPSE mesurement using M mode in the deep transgastric right heart view at zero degrees

CONTACTS AND LOCATIONS:
Overall Officials: Lalitha Manickam, Principal Investigator — NUH
Locations (1):
- National university Hospital, Singapore, Singapore